CLINICAL TRIAL: NCT01899989
Title: Stereotactic Body Radiation Therapy for Inoperable Locally-advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-113
Record Dates: First submitted 2013-07-08; First posted 2013-07-16 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stereotactic Body Radiation Therapy (SBRT); Chemotherapy; 13-113
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A) >5cm,Chemo eligible (closed to accrual) (Experimental): Patients will receive five fractions of either 8, 10, or 12 Gy to the gross tumor only. Following SBRT patients will be evaluated by their medical oncologist for consideration of adjuvant chemotherapy, starting 6-8 weeks post-RT. All patients will be followed for one year. Patients will be assessed for toxicity by their radiation oncologist at 4 to 6 weeks post-RT and during chemotherapy by their medical oncologist. Follow up after completion of all treatment will consist of CT chest scans at 6 and 12 months post-SBRT and toxicity assessments every 3 months from the end of SBRT for one year.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: cisplatin or carboplatin-based
- B) 3-5cm OR Chemo ineligible (Experimental): Using intensity-modulated radiation therapy (IMRT) or volumetric arc therapy (VMAT), the choice of which is determined by the radiation oncologist, patients will be treated in < 5 fractions every other day. The total treatment dose will be between 45 and 54 Gy in < 5 fractions per standard of care. All patients will be followed for one year. Patients will be assessed for toxicity by their radiation oncologist at 4 to 6 weeks post-RT and during chemotherapy at the discretion of their medical oncologist. Follow up after completion of all treatment will consist of CT chest scans at 6 and 12 months post-SBRT and toxicity assessments every 3 months from the end of SBRT for one year. FDG PET/CT scans and Pulmonary Function Tests (PFTs) will be obtained at 3 months and 9 months after SBRT.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT)
Drug: cisplatin or carboplatin-based — Standard chemotherapy with a histology-selected cisplatin or carboplatin-based doublet will be administered intravenously as adjuvant therapy. Gemcitabine will be used for squamous cell carcinomas and pemetrexed will be used for non-squamous non-small cell lung cancer. Cisplatin or carboplatin will be used in combination with the histology-selected agent. The choice of cisplatin or carboplatin will be at the discretion of the treating medical oncologist.
  Arms: A) >5cm,Chemo eligible (closed to accrual)

SUMMARY:
The purpose of this study is to determine if the use of exploratory immunologic biomarkers, functional MRI images can serve as early predictors for response of NSCLC. It also will provide important information on the perceived side effects from a patient perspective. Patients may participate if they have tumors ≥3 cm without lymph node involvement (for which chemotherapy is not part of the standard of care). Patients will only receive stereotactic body radiation therapy (SBRT) per standard dose guidelines.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Histologically confirmed non-small cell lung cancer
* Medically or technically inoperable as per thoracic surgeon or patient's preference not to undergo surgical resection
* Age ≥ 18 years
* Women of childbearing potential must have a negative blood pregnancy test
* Ability to provide written informed consent

Cohort A:

* Stage IIA-IIIA (TanyN1M0 or T2b-4N0M0) Selected patients with single station N2 nodal involvement in close proximity to the primary tumor target may be considered eligible at the discretion of the PI if all normal tissue guidelines can be met
* Eligible for chemo-therapy
* Karnofsky Performance Status ≥70%
* Men and women of childbearing potential must be willing to use effective contraception while on treatment and for at least 3 months thereafter
* Patients must show adequate organ function as defined by:

  * Calculated creatinine clearance ≥40 mL/min for patients receiving pemetrexed (by Cockcroft-Gault)
  * Calculated creatinine clearance ≥30 mL/min for patients receiving gemcitabine or paclitaxel (by Cockcroft-Gault) Total bilirubin less than 1.5 x ULN (unless known Gilbert's disease)
  * AST and ALT less than 3 x ULN
  * Absolute neutrophil count greater than 1500/mm3
  * Platelet count greater than 100,000/mm3

Cohort B:

* T2a-4N0M0 who are not candidates for cohort A or who will not be treated with chemotherapy (due to patient preference or at the recommendation of the treating physician).

Exclusion Criteria:

All patients:

* Prior radiation therapy to the lungs
* Prior surgery or chemotherapy for this presentation of lung cancer (history of prior lung cancer that has been treated and deemed inactive by the clinician is acceptable. Recurrent tumors may be treated on protocol as long as SBRT will be the definitive treatment.)
* N2-3 lymph node involvement based on PET/EBUS-FNA/mediastinoscopy (Any N2 disease that is more than just minimal single station involvement is excluded)
* Direct tumor extension into including aorta or pulmonary artery
* Chronic corticosteroid use equivalent to ≥ prednisone 10 mg daily

Prior treatment with a CD137 agonist, ipilimumab, or the CTLA-4 inhibitor, or PD-1/PDL-1 inhibitor

* Unstable congestive heart failure

Cohort A:

* Continuous oxygen use

Patients meeting the following exclusion criteria will be excluded from the functional MRI portion only:

* Metallic implant,exclusions will be determined per institutional policies
* Pacemaker and defibrillators are excluded
* Stents etc. will be evaluated according to MSKCC policy
* Unmanageable claustrophobia
* High risk for nephrogenic systemic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-07-05 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (Cohort A) | 2 years
  standard 3+3 dose-escalation scheme

SECONDARY OUTCOMES:
≥ grade 4 or persistent ≥ grade 3 late toxicities (Cohorts A & B) | ≥3 months post SBRT
  All patients will be assessed for toxicities according to CTCAE v 4.0 at least once during SBRT.
overall survival (Cohorts A & B) | 2 years
  Response and progression will be evaluated per standard of care for radiographic progression on CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Wu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/